CLINICAL TRIAL: NCT02638298
Title: Incisional Negative Pressure Wound Therapy for Preoperatively Irradiated Lower Extremity Soft Tissue Sarcoma Wounds. A Prospective Randomized Clinical Trial
Brief Title: Incisional Negative Pressure Wound Therapy for Preoperatively Irradiated Lower Extremity Soft Tissue Sarcoma Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00028423
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Cancer; Infectious Disease
MeSH Terms: conditions — Sarcoma; Neoplasms; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPWT dressing (Experimental)
  Interventions: Device: Prevana Dressing
- Standard dry gauze dressing (Placebo Comparator)
  Interventions: Other: Standard Dry Gauze Dressing

INTERVENTIONS:
Device: Prevana Dressing — negative pressure wound therapy (NPWT) dressing
  Arms: NPWT dressing
Other: Standard Dry Gauze Dressing — Standard Dry Gauze Dressing
  Arms: Standard dry gauze dressing

SUMMARY:
This is a study comparing two methods of dressing a post operative wound that are currently in practice. One method is a traditional dry gauze dressing. The other method is using a negative pressure dressing that provides gentle suction on the wound.

The investigators will attempt to determine how well the use of post-operative negative pressure dressing reduces wound healing problems in patients who have surgery after radiation for a sarcoma in the thigh or leg.

DETAILED DESCRIPTION:
Postoperative surgical site infections pose a significant challenge to the orthopaedic oncologist, especially in wounds that have been previously irradiated with neo adjuvant external beam radiation therapy (EBRT). There are many studies demonstrating the relatively high risk of wound complications after lower extremity sarcoma resection. Published data suggest that these preoperatively radiated wounds have a postoperative infection rate of 17%-44% with "traditional" dressings (e.g. dry gauze surgical dressings).

A prospective series of 190 patients and showed a wound complication risk of 35% in preoperative irradiated wounds. The morbidity associated with wound complications can range from moderate (prolonged dressing changes) to severe (life or limb threatening infection). Patients who develop wound complications have been shown to longer hospitalizations and higher costs [ref]. Anatomic location of the tumor has been shown to be a risk factor for the development of wound complications with lower extremities being higher risk than upper extremities. There are several published studies examining the effect of negative pressure wound therapy (NPWT) on high risk surgical wounds. Abdominal wound complications can be reduced with the use of incisional NPWT. In the orthopaedic literature the use of negative pressure incisional dressings have been shown to lower the risk of wound complications in total hip arthroplasty, acetabular fractures, and extremity fractures.

To our knowledge, there have not been any published studies on the utility of negative pressure wound therapy in previously irradiated soft tissue sarcoma wounds. The investigators feel that this high risk patient cohort could potentially benefit from reducing wound complications through NPWT and is an ideal population to study its effect.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Willing to consent to randomization and able to participate in the study
* Lower extremity soft tissue sarcoma necessitating radiation prior to surgical resection
* Primary closure of wound
* Patients scheduled for surgical resection

Exclusion Criteria:

* Flap coverage or skin graft
* Patients scheduled for amputations as local control of their tumor
* Sarcomas where radiation is not planned preoperatively
* Repeat surgeries for oncologic reasons (positive margins)
* Known allergy to adhesive tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee R Leddy, MD, Principal Investigator — Medical University of South Carolins
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data safety and monitoring will be provided by the Hollings Cancer Center DSMC. This committee will serve for all sites. The DSMC meets 6 times a year and reviews all MUSC IRB adverse events, protocol deviations/violations, early stopping rules and internal audit results. The PI will be responsible for identifying, reviewing monthly, and reporting adverse events.
  Individual participant data will not be shared between the sites. All data will be deidentified and linked with a code.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to NPWT or dry gauze dressing following oncologic resection and were excluded in the settings of amputation, revision, or flap coverage
Period: Overall Study
Arm/Group | NPWT Dressing | Standard Dry Gauze Dressing
Started | 81 | 79
Completed | 81 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for sex of participants.
Groups:
- NPWT Dressing: Prevana Dressing: negative pressure wound therapy (NPWT) dressing. Baseline characteristics were not collected for sex of participants, nor was the age documented as a result of all participants being over the age of 18.
- Standard Dry Gauze Dressing: Standard Dry Gauze Dressing: Standard Dry Gauze Dressing. Baseline characteristics were not collected for sex of participants, nor was the age documented as a result of all participants being over the age of 18.
- Total: Total of all reporting groups
Arm/Group | NPWT Dressing | Standard Dry Gauze Dressing | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Customized [Count of Participants; unit: Participants]
  >=18 years old | 81 | 79 | 160
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data were not collected and therefore, sex-specific analyses of baseline characteristics and outcomes cannot be performed.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Wound Complication Rate
Description: To estimate the wound complication rate of post-operative negative pressure dressings and traditional dry dressings, and risk of secondary interventions after resection of soft tissue sarcoma in lower extremities that have received pre-operative radiation.
  Post-operative pain severity assessed by Visual analogue scale at 2 weeks and 6 months post-operatively where visual analogue scale ranges from zero to ten where (0 = no pain, 10 = maximum pain imaginable).
Time Frame: longitudinally up to 6 months postoperatively
Population: Post-operative pain severity assessed by Visual analogue scale at 2 weeks and 6 months post-operatively where visual analogue scale ranges from zero to ten where (0 = no pain, 10 = maximum pain imaginable).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NPWT Dressing | Standard Dry Gauze Dressing
Number analyzed (Participants) | 81 | 79
score on a scale
  Post-operative pain severity assessed by Visual analogue scale at 2 weeks postoperatively. | 3.7 (2.2) | 3.7 (2.5)
  Post-operative pain severity assessed by Visual analogue scale at 6 months postoperatively. | 2.1 (1.9) | 2.2 (1.9)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | NPWT Dressing | Standard Dry Gauze Dressing
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 0/81 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02638298/Prot_SAP_000.pdf